CLINICAL TRIAL: NCT07043582
Title: Tinea Capitis Patients: The Predictive Value of Trichoscopic Findings for Treatment Response - A Prospective Observational Study
Brief Title: Trichoscopic Predictors of Treatment Response in Tinea Capitis: A Prospective Study
Acronym: TCTREP
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Tunç Ozen, Principal Investigator, Istanbul Medeniyet University
Other Study IDs: 2536854
Record Dates: First submitted 2025-05-23; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Tinea Capitis
Keywords: tinea capitis; dermotoscopy; trichoscopy; wood lamp; mycology
MeSH Terms: conditions — Tinea Capitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Hair shafts, scalp scales, and fungal cultures obtained from affected areas will be retained for microbiological analyses, including potassium hydroxide (KOH) examination, fungal culture, species identification, and MALDI-TOF MS analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brief Summary (Plain Language Version)

The goal of this observational study is to learn how well changes seen under a special microscope called a trichoscope (used to look at hair and scalp) match the success of treatment in children and adolescents with a scalp fungal infection called tinea capitis. The main questions it aims to answer are:

Do changes in trichoscopic findings show when the fungal infection is cured?

Does having more severe trichoscopic findings at the start mean that treatment will take longer or be less successful?

Do different fungus types respond differently to the same treatment?

Participants will:

Be between the ages of 0 and 18 with confirmed tinea capitis based on lab tests (microscopy and/or culture)

Receive an oral antifungal medicine called terbinafine for 4 weeks (dosing based on weight)

Attend regular checkups every 4 weeks until both scalp appearance and lab tests show the infection is gone

At each visit, participants will:

Have their scalp examined using a trichoscope

Provide scalp samples for fungal testing

Be assessed for symptoms like itching, redness, and scaling

The study will also look at how fast different signs on the scalp go away, and which of these signs are best at predicting whether the fungus is still present.

DETAILED DESCRIPTION:
This prospective observational study aims to evaluate the predictive value of trichoscopic findings for treatment response in pediatric patients (ages 0-18) diagnosed with tinea capitis. Tinea capitis is a fungal infection of the scalp that commonly affects children. Diagnosis will be confirmed through clinical evaluation, dermoscopic examination, and laboratory testing, including potassium hydroxide (KOH) smear and fungal culture from scalp samples. Only patients with laboratory-confirmed tinea capitis (positive KOH and/or culture) will be enrolled.

The primary objective is to determine the correlation between trichoscopic changes and mycological cure, defined as both KOH and culture negativity following systemic antifungal treatment with terbinafine. Secondary objectives include evaluating the timeline of regression for individual trichoscopic signs, determining whether certain dermoscopic features persist despite microbiological cure, and assessing whether specific patterns are predictive of treatment resistance. Additionally, the study aims to investigate if baseline trichoscopic scores or fungal species (e.g., Microsporum canis, Trichophyton tonsurans, T. violaceum) are associated with prolonged treatment duration or lower cure rates.

Eligible patients will receive weight-adjusted oral terbinafine therapy for four weeks and return for clinical, trichoscopic, and microbiological evaluation every four weeks thereafter until both clinical and mycological cure are achieved. At each follow-up, standardized data will be collected including clinical symptoms (e.g., erythema, scaling, hair loss), trichoscopic features (e.g., comma hairs, corkscrew hairs, black dots), and laboratory results. Trichoscopic evaluations will be recorded using handheld dermoscopy and interpreted independently by two dermatologists. Discrepancies will be resolved by a third expert reviewer.

Statistical analyses will include descriptive statistics, McNemar's test to assess pre/post-treatment trichoscopic changes, sensitivity/specificity/PPV/NPV analyses for predicting culture positivity, and Kaplan-Meier survival analysis for the regression timing of individual dermoscopic findings. Regression models will explore predictors of treatment duration and failure. A trichoscopic scoring system will also be evaluated as a tool for estimating treatment response.

All procedures will comply with the Declaration of Helsinki, and written informed consent will be obtained from legal guardians. Patient confidentiality will be maintained throughout the study. The findings are expected to enhance early treatment monitoring and guide clinical decisions using non-invasive imaging tools.

ELIGIBILITY:
Inclusion Criteria:

* Age between 0 and 18 years

Clinical and trichoscopic findings compatible with tinea capitis

Laboratory confirmation of tinea capitis (positive potassium hydroxide [KOH] smear and/or fungal culture)

Eligible for systemic antifungal treatment with terbinafine

Written informed consent obtained from a parent or legal guardian

Exclusion Criteria:

* Age over 18 years

Negative KOH smear and negative culture

Current use of immunosuppressive therapy or presence of severe systemic illness (e.g., malignancy, HIV, organ transplant)

Contraindication to terbinafine treatment

Poor compliance or unwillingness to attend follow-up visits

Coexisting dermatologic conditions in the affected scalp area (e.g., seborrheic dermatitis, alopecia areata, lichen planus)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of pediatric patients aged 0 to 18 years with clinically and dermoscopically suspected tinea capitis, confirmed by potassium hydroxide (KOH) smear and/or fungal culture. Participants are recruited from dermatology outpatient clinics and must be eligible for systemic antifungal treatment. The study focuses on this age group as tinea capitis primarily affects children and adolescents.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-07-24 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with disappearance of characteristic trichoscopic findings at the time of mycological cure | Up to 12 weeks (until mycological cure is achieved)
  The primary outcome is the proportion (%) of patients who exhibit complete regression of characteristic trichoscopic findings (e.g., black dots, comma hairs, corkscrew hairs) as assessed by trichoscopic examination, at the time of mycological cure. Mycological cure is defined as negative results on both potassium hydroxide (KOH) smear and fungal culture.

CONTACTS AND LOCATIONS:
Overall Officials: Vefa Aslı Erdemir, Proffesor, Study Director — medeniyet university
Locations (1):
- Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No